CLINICAL TRIAL: NCT04410159
Title: A Pilot, Open-Labelled, Randomised Controlled Trial Of Povidone-Iodine Vs Essential Oil And Tap Water Gargling For COVID-19 Patients
Brief Title: Povidone-Iodine Vs Essential Oil Vs Tap Water Gargling For COVID-19 Patients
Acronym: GARGLES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universiti Sains Islam Malaysia (Other)
Collaborators: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, NURUL AZMAWATI MOHAMED, Dr, Universiti Sains Islam Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USIMalaysia
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: gargle; povidone-iodine; essential oils; tap water
MeSH Terms: conditions — COVID-19 | interventions — Povidone-Iodine; Oils, Volatile; Listerine

STUDY DESIGN:
Intervention Model Description: 4 arms
  1. Gargle with povidone-iodine
  2. Gargle with essential oils
  3. Gargle with tap water
  4. Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Povidone-iodine (Experimental): gargle with povidone-iodine 10mL, 30 seconds, 3 times per day, 7 days
  Interventions: Drug: Povidone-Iodine
- Essential Oils (Experimental): gargle with essential oils 20mL, 30 seconds, 3 times per day, 7 days
  Interventions: Drug: Essential oils
- Tap water (Experimental): gargle with tap water 100 mL, 30 seconds, 3 times per day, 7 days
  Interventions: Other: Tap water
- Control (No Intervention): This group will receive the standard treatment protocol without any additional intervention

INTERVENTIONS:
Drug: Povidone-Iodine — Gargle
  Other Names: Betadine
  Arms: Povidone-iodine
Drug: Essential oils — Gargle
  Other Names: Listerine
  Arms: Essential Oils
Other: Tap water — Gargle
  Arms: Tap water

SUMMARY:
The purpose of this study is to assess the ability of regular gargling to eliminate severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in the throat and nasopharynx. This 4 arms interventional study compares the effect of gargling using povidone-iodine, essential oils- based, tap water with control (no intervention) among Stage 1 coronavirus disease-2019 (COVID-19) patients.

Findings from this study will provide new insight into the importance of gargling in the treatment and prevention of COVID-19.

DETAILED DESCRIPTION:
Experimental plan

After consent is taken, all groups will be briefed regarding the study protocol separately.

* Group A will be briefed on the correct procedures of gargling with Betadine®. The participants will be instructed to take 10ml of povidone-iodine (PVP-I), tilt their heads backward and gargle for 30 seconds, three times per day for 7 days
* Group B will be briefed on the correct technique of gargling with Listerine®. The participants will be instructed to take 20ml of essential oils, tilt their heads backward and gargle for 30 seconds, three times per day for 7 days
* Group C will be briefed on the correct technique of gargling with hydrogen peroxide. The participants will be instructed to take 10ml of hydrogen peroxide, tilt their heads backward and gargle for 30 seconds, three times per day for 7 days
* Group D will be briefed about the involvement in this study. They will be managed according to the standard protocol of the hospital with no additional intervention.

Monitoring

1. Oropharyngeal and nasopharyngeal swabs will be taken on day 4, 6 of intervention, and day 12 post-intervention. The swabs will be subjected to detection of SARS-CoV-2 by real-time reverse transcriptase-polymerase chain reaction (rt RT-PCR).
2. Patients will be given a chart for them to record their gargling practice and symptoms (if any) during the intervention period ( 7 days)
3. Clinical data collection sheet will be provided to attending clinicians. The required information includes demographic data, daily vital signs, serial absolute lymphocytic count, LDH, chest radiograph, and symptoms. Clinical monitoring will be done until day 14 of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. adult aged 18 years and above
2. able to understand instructions
3. Stage 1 COVID-19
4. < 5 days of illness or diagnosis

Exclusion Criteria:

1. Less than 18 years old
2. Unable to understand instructions
3. Stage 2 & 3 COVID-19
4. Respiratory symptoms or fever on admission
5. Abnormal chest radiograph or computed tomography (CT) findings on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NURUL A MOHAMED, Principal Investigator — Universiti Sains Islam Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Bandar Tun Razak, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The participant data from the final research dataset used in the published manuscript will be shared upon reasonable request. The protocol and data analysis will be shared in clinicaltrial
Supporting Information: Study Protocol, ICF
Time Frame: September to December 2020
Access Criteria: email to drnurul@usim.edu.my

REFERENCES:
- [Background] Eggers M, Koburger-Janssen T, Eickmann M, Zorn J. In Vitro Bactericidal and Virucidal Efficacy of Povidone-Iodine Gargle/Mouthwash Against Respiratory and Oral Tract Pathogens. Infect Dis Ther. 2018 Jun;7(2):249-259. doi: 10.1007/s40121-018-0200-7. Epub 2018 Apr 9. PMID 29633177
- [Background] Eggers M. Infectious Disease Management and Control with Povidone Iodine. Infect Dis Ther. 2019 Dec;8(4):581-593. doi: 10.1007/s40121-019-00260-x. Epub 2019 Aug 14. PMID 31414403
- [Background] Dennison DK, Meredith GM, Shillitoe EJ, Caffesse RG. The antiviral spectrum of Listerine antiseptic. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1995 Apr;79(4):442-8. doi: 10.1016/s1079-2104(05)80124-6. PMID 7614202
- [Background] Satomura K, Kitamura T, Kawamura T, Shimbo T, Watanabe M, Kamei M, Takano Y, Tamakoshi A; Great Cold Investigators-I. Prevention of upper respiratory tract infections by gargling: a randomized trial. Am J Prev Med. 2005 Nov;29(4):302-7. doi: 10.1016/j.amepre.2005.06.013. PMID 16242593

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited 2 to 3 days after date of diagnosis (nasophryngeal swab postive for SARS-C0V-2. All patients were asymptomatic and admitted to the hospital for observation
Pre-assignment Details: No significant event occurred after enrollment
Period: Overall Study
Arm/Group | Povidone-iodine | Essential Oils | Tap Water | Control
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: This group received the standard treatment protocol without any additional intervention
- Total: Total of all reporting groups
Arm/Group | Povidone-iodine | Essential Oils | Tap Water | Control | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (7.44) | 34.4 (12.50) | 30.8 (3.77) | 24.8 (2.68) | 30.6 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 0 | 4
  Male | 2 | 4 | 5 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 5 | 5 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malaysia | 5 | 5 | 5 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Early Viral Clearance
Description: Viral clearance is defined as two negative RT-PCR (of swabs from oropharynx and nasopharynx) results at least 24 hours apart
Time Frame: Day 6
Measure: Count of Participants; unit: Participants
Arm/Group | Povidone-iodine | Essential Oils | Tap Water | Control
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 5 | 4 | 1 | 0

2. Secondary Outcome: Number of Participants With Negative RT-PCR Results
Description: RT-PCR (swabs from oropharynx and nasopharynx) taken at day 12
Time Frame: Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | Povidone-iodine | Essential Oils | Tap Water | Control
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 5 | 4 | 2 | 1

3. Secondary Outcome: Number of Patients That Progress to More Severe Disease
Description: Presence of signs and symptoms of more severe COVID19 Based symptoms diary and clinical evaluation
Time Frame: Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | Povidone-iodine | Essential Oils | Tap Water | Control
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Patients With Abnormal Radiological Findings
Description: abnormal chest x-ray or CT scan
Time Frame: Day 0-14
Measure: Count of Participants; unit: Participants
Arm/Group | Povidone-iodine | Essential Oils | Tap Water | Control
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Abnormal Laboratory Findings
Description: Abnormal absolute lymphocytic count Abnormal C-reactive protein
Time Frame: Day 0-14
Measure: Count of Participants; unit: Participants
Arm/Group | Povidone-iodine | Essential Oils | Tap Water | Control
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from day 1 of intervention until day 14
Description: Similar to clinicaltrial.gov
Arm/Group | Povidone-iodine | Essential Oils | Tap Water | Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Inadequate budget for laboratory test lead to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT04410159/Prot_SAP_ICF_000.pdf